CLINICAL TRIAL: NCT05671848
Title: Study of the Activity of the Ventral Intermediate Nucleus of the Thalamus Under Ecological Conditions in Essential Tremor.
Brief Title: Electroclinical Correlates in Essential Tremor
Acronym: ECOLOVIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Collaborators: MINDig (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2022/29
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Essential Tremor
Keywords: Essential Tremor; Local field potentials; Deep Brain Stimulation
MeSH Terms: conditions — Essential Tremor

STUDY DESIGN:
Intervention Model Description: Single-center, open-label, prospective cohort pilot study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- experimental arm (Experimental): Patient with ET and Receiving deep brain stimulation treatment with implantation of the PERCEPT™ device
  Interventions: Other: Recordings of thalamic activity

INTERVENTIONS:
Other: Recordings of thalamic activity — Recordings of thalamic activity will be performed at home, in ecological conditions. They will be realized during 4 distinct conditions each week between M3 and M6 post implantation: at rest and during tremor-induced movements. For these recordings, stimulation will be either turned Off or On. Three successive recordings of 30 seconds separated by 1 minute will be made for each condition.

SUMMARY:
Essential tremor (ET) is a neurological disorder that affects nearly 0.9% of the world's population. High-frequency Deep Brain Stimulation (DBS) of the ventral-intermediate nuclei of the thalamus (VIM) has been proven as an effective second-line treatment for severe forms of ET.

The arrival on the market of the PERCEPT™ (new stimulator/recorder, Medtronic, Minneapolis, USA) now allows, in addition to the stimulation delivery, the recording of intracerebral activity at a distance from surgery, in a non-invasive way and in ecological condition at home. Investigators aim at recording the variations of thalamic Local Field Potentials (LFP) oscillations, in ecological condition, during rest and movement, with and without deep brain stimulation, once a week, between M3 and M6 post surgery.

DETAILED DESCRIPTION:
Essential tremor (ET) is a neurological disorder that affects nearly 0.9% of the world's population, including 300,000 people in France alone. Patients who suffer from this condition usually present an upper limb tremor during voluntary motor activities but not at rest. The pharmacological treatments proposed for this condition are only effective in about 50% of patients, and this effectiveness is often only partial or observed at the cost of unacceptable side effects. Since the end of the 1980's, high-frequency deep brain stimulation (DBS) of the ventral-intermediate nuclei of the thalamus (VIM) has been proposed as an effective second-line treatment for severe forms of ET. However, some neuro-stimulated patients experience a recurrence of their tremor and may complain of an increase in pre-existing cerebellar ataxia. The mechanisms underlying these phenomena are still debated, but the fact that VIM stimulation is applied in a chronic and undifferentiated manner seems to play a determining role. One way to circumvent these phenomena could be to stimulate the VIM only during movement since the tremor in this condition is an action or postural tremor. This type of "closed-loop therapy" requires one or more intracerebral tremor biomarkers that can be reliably recognized and used to automatically trigger or modulate the intensity of VIM stimulation only when necessary. In a preliminary study in 10 patients, the investigators of Bordeaux university hospital were able to demonstrate the existence of potential intracerebral biomarkers of tremor under experimental conditions,in the immediate postoperative period (Guehl et al. 2022, submitted). The arrival on the market of the PERCEPT™ (new stimulator/recorder, Medtronic, Minneapolis, USA) now allows, in addition to treating patients with DBS, the recording of intracerebral activity at a distance from surgery, in a non-invasive way and in ecological condition at home. This study aim at recording the variations of thalamic oscillations, in ecological condition, during rest and movement, with and without deep brain stimulation. These measurements will be performed once a week during the 12 weeks of the late post-operative period (from 3 to 6 months), in order to ensure the reproducibility of the results. The signal processing and analysis will be performed in a blind manner to the patient's activity and stimulation condition.

ELIGIBILITY:
Inclusion Criteria:

* Advanced disabling and drug-resistant tremor
* Receiving deep brain stimulation treatment with implantation of the PERCEPT™ device according to standard care
* Chronic progressive cardiac, renal, hematological or pulmonary diseases under treatment.
* Patient aged between 18 to 75 years
* Normal brain MRI
* MATTIS score ≥ 130/144 or MOCA ≥ 24/30
* Subject affiliated with or benefiting from a social security plan
* Free, informed and written consent signed by the participant and the investigator (at the latest on the day of inclusion and before any examination required by the research)

Exclusion Criteria:

* Major depressive syndrome (Beck scale > 20)
* MRI showing significant brain atrophy or significant hypersignals
* Pregnant or breastfeeding women
* Being unable to give personal consent
* Be subject to a measure of legal protection (curatorship, guardianship) or placed under judicial protection.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2023-05-03 (Actual); Primary Completion 2026-05-03 (Estimated); Study Completion 2026-05-03 (Estimated)

PRIMARY OUTCOMES:
Recorded signal quality | 6 months (M6) after surgery (M0)
  The primary endpoint of this study will be the recorded signal quality, i.e., the ratio of signal amplitude (thalamic oscillations) to noise (artifacts) at least 3/1.

SECONDARY OUTCOMES:
presence or absence of brain oscillations | 6 months (M6) after surgery (M0)
  Good reproducibility of the electrical signals based on the ability to visually individualize, from successive recordings, the presence or absence of brain oscillations in the different frequency bands of interest (peaks on the power spectrum). For this purpose, the intra-patient reproducibility of the spectral powers at rest and in activity will be estimated using Cohen's Kappa coefficient and its two-sided 95% confidence interval according to the exact binomial law.
Power spectral density (PSD) | 6 months (M6) after surgery (M0)
  Analysis of the amplitude of the average PSDs in the 2 distinct motor conditions (rest/movement) and in the 2 stimulation conditions (inactive/active). A difference in PSD amplitude of 15% between the 4 situations is necessary to conclude to significant differences.
Location of the electrodes | 1 month (M1) after surgery (M0)
  Position of the electrodes and the contacts used for the LFP recordings will be analyzed. These contacts will need to be positioned in each VIM that are the targets of deep brain stimulation in the ET.
Evaluation of the efficacy of VIM DBS in the ET | 3 months (M3) after surgery (M0)
  A 50% reduction in clinical scores at M3 compared to the pre-operative scores (M-1) is necessary to conclude that deep brain stimulation of VIM is significantly effective on tremor.

CONTACTS AND LOCATIONS:
Overall Officials: Dominique GUELH, Pr, Study Director — University Hospital, Bordeaux; Edouard COURTIN, Dr, Principal Investigator — University Hospital, Bordeaux; Mahmoud HASSAN, Dr, Study Chair — MINDig
Locations (1):
- CHU de Bordeaux, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No